CLINICAL TRIAL: NCT00878683
Title: Exploring the Use of a Novel Device for Reducing Catheter-Related Bloodstream Infections
Brief Title: Novel Device for Reducing Catheter-Related Infections
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never received IRB approval; Withdrawn before enrollment ever started
Sponsor: University of Kansas (Other)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Stephen Waller MD, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11525
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Intensive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Device and standard catheter
  Interventions: Device: silicone catheter boot
- 2 (No Intervention): Standard catheter

INTERVENTIONS:
Device: silicone catheter boot — silicone device using Dermabond
  Arms: 1

SUMMARY:
This study is a pilot study of the safety, tolerability and efficacy of an investigational central venous catheter device used in conjunction with a standard central venous catheter. The hypothesis is that utilization of a catheter device incorporating cyanoacrylate will reduce catheter colonization by bacteria, and may decrease the rate of catheter-related bloodstream infections.

ELIGIBILITY:
Inclusion Criteria:

* Admission in the ICU at time of catheter insertion
* Indication for central venous catheter placement
* De novo catheter insertion in the subclavian or internal jugular veins

Exclusion Criteria:

* Anticipated catheter duration < 72 hours
* Planned guidewire exchange
* Documented bacteremia within 48 hours prior to catheter placement
* Extensive skin breakdown near the site of potential catheter placement
* Emergent line placement
* Screening labs with ANC < 500 or platelets < 50K
* Hypersensitivity to cyanoacrylates or formaldehyde
* Prior enrollment in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Catheter site inspection | Baseline, Daily

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Waller, MD, Principal Investigator — University of Kansas Medical Center